CLINICAL TRIAL: NCT04774952
Title: A Phase 1/1b, Open-Label, Multicenter, Dose-Escalation Study of RMC 5552 Monotherapy in Adult Subjects With Relapsed/Refractory Solid Tumors
Brief Title: Dose Escalation of RMC-5552 Monotherapy in Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-5552-001
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors
Keywords: PIK3CA; PTEN; TSC1/2; STK11; MTOR; MYC; MAPK; advanced solid tumor; advanced solid malignancies; melanoma; skin cancer; ovarian cancer; endometrium/uterus cancer; bladder cancer; cervical cancer; Carcinoma, Non-Small-Cell Lung; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Esophageal Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Neoplasms, Glandular and Epithelial; Gastrointestinal Neoplasms; Digestive System Neoplasms; Head and Neck Neoplasms; Digestive System Diseases; Esophageal Diseases; Gastrointestinal Diseases; 4EBP1
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Melanoma; Skin Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Esophageal Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Neoplasms, Glandular and Epithelial; Gastrointestinal Neoplasms; Digestive System Neoplasms; Head and Neck Neoplasms; Digestive System Diseases; Esophageal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RMC-5552 (Experimental): RMC-5552 for IV administration
  Interventions: Drug: RMC-5552

INTERVENTIONS:
Drug: RMC-5552 — RMC-5552 for IV administration

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) profiles of escalating doses of RMC-5552 monotherapy in adult participants with relapsed/refractory solid tumors and to identify the recommended Phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of RMC-5552 monotherapy in participants with advanced relapsed or refractory solid tumors. The study will include 2 components: 1) a Dose-Escalation Component for participants with relapsed or refractory solid tumors and 2) a Dose-Expansion Component for participants with relapsed or refractory solid tumors harboring certain specific mutations/rearrangements that result in hyperactivation of the mTOR pathway. Participants will be treated until disease progression per RECIST v1.1, unacceptable toxicity, or other criteria for withdrawal are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants (male or female) ≥18 years of age
* Participants who have advanced solid tumors that have failed, are intolerant to, or are considered ineligible for standard of care anticancer treatments including approved drugs for oncogenic drivers in their tumor type
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participants in the Dose-Expansion Component must have molecular aberrations in the mTOR pathway
* Adequate hematologic, hepatic and renal function

Exclusion Criteria:

* Known or suspected leptomeningeal or brain metastases or spinal cord compression
* Primary central nervous system (CNS) tumors
* Clinically significant cardiac disease
* Active, clinically significant interstitial lung disease or pneumonitis
* Subjects with abnormal fasting glucose, type 1 diabetes, or uncontrolled type 2 diabetes are excluded.
* Subjects with stomatitis or mucositis of any grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | up to 3 years
  Incidence, nature, and severity of treatment-emergent AEs and serious AEs, including incidence and severity of findings in laboratory values or vital signs for RMC-5552 monotherapy
Number of participants with dose limiting toxicities (DLTs) | 21 days
  Incidence and nature of DLTs with RMC-5552 monotherapy

SECONDARY OUTCOMES:
Cmax | up to 3 years
  Peak plasma concentration of RMC-5552
Tmax | up to 3 years
  Time to achieve peak plasma concentration of RMC-5552
Area Under the Curve (AUC) | up to 3 years
  Area under the plasma concentration time curve of RMC-5552
t1/2 | up to 3 years
  Elimination half-life of RMC-5552
Accumulation Ratio | up to 3 years
  Ratio of accumulation of RMC-5552 from a single dose to steady state with repeated dosing
Overall Response Rate (ORR) | up to 3 years
  Overall response rate of RMC-5552 per RECIST v1.1
Duration of Response (DOR) | up to 3 years
  Duration of response of RMC-5552 per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc, Study Director — Revolution Medicines, Inc.
Locations (8):
- United States (8):
  - UC Irvine - Chao Family Comprehensive Cancer Center, Irvine, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Dell Seton Medical Center at University of Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schram AM, Naqash AR, Haura EB, Riess JW, Ulahannan SV, Ou SI, Munster PN, Cheng ML, Gustafson WC, Bitman B, Friedman R, Penn R, Kar S, Seshadri V, Wang Z, Tao L, Yang YC, Singh M, Burris HA, Meyerowitz JG. The Bi-steric, mTORC1-Selective Inhibitor, RMC-5552, in Advanced Solid Tumors: A Phase 1 Trial. Clin Cancer Res. 2025 Dec 1;31(23):4933-4943. doi: 10.1158/1078-0432.CCR-25-2112. PMID 41056387